CLINICAL TRIAL: NCT06466525
Title: A Two-Part Single and Multiple Ascending Dose Trial of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LBT-3627 in Healthy Participants and in Participants With Parkinson's Disease.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Longevity Biotech Australia Pty Ltd (subsidiary) (Industry)
Responsible Party: Sponsor
Organization: Longevity Biotech (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBT-3627-101
Record Dates: First submitted 2024-06-10; First posted 2024-06-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — LBT-3627

STUDY DESIGN:
Intervention Model Description: Placebo controlled, double blind, SAD and MAD dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled, double blind (patient and investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteers - SAD (Experimental): Single dose of LBT-3627 administered to healthy volunteers
  Interventions: Drug: LBT-3627; Drug: Placebo
- Parkinson's disease patients - SAD (Experimental): Single dose of LBT-3627 administered to Parkinson's disease patients
  Interventions: Drug: LBT-3627; Drug: Placebo
- Parkinson's disease patients - MAD (Experimental): Multiple doses of LBT-3627 administered to Parkinson's disease patients
  Interventions: Drug: LBT-3627; Drug: Placebo

INTERVENTIONS:
Drug: LBT-3627 — Synthetic peptide
Drug: Placebo — Vehicle

SUMMARY:
Phase I a/b SAD/MAD study to evaluate safety and tolerability of LBT-3627 in both healthy volunteers and Parkinson's patients.

DETAILED DESCRIPTION:
Evaluate the safety and tolerability of LBT-3627 in both a single and multiple ascending dose study.

Phase Ia will explore safety and tolerability first in healthy volunteers then followed by Parkinson's patients after a single dose. Dose levels will escalate per cohort.

Phase Ib will explore safety and tolerability in Parkinson's patients after multiple doses. Dose levels will escalate per cohort.

ELIGIBILITY:
Inclusion Criteria (Everyone)

Participants will be included in the study only if they satisfy all the following criteria:

1. Must have given written informed consent, before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Healthy male or female, aged between 30 and 89 years, inclusive at screening.
3. Body mass index (BMI) of 18 to 32 kg/m2, inclusive.
4. Physical examination without any additional clinically relevant findings
5. Systolic blood pressure in the range of 90 to 140 mmHg (inclusive) and diastolic blood pressure in the range of 40 to 90 (inclusive) mmHg after 5 minutes in supine/semi-supine, and subsequently after 3 minutes of standing position.

   Note 1: Participants with orthostatic hypotension are not permitted. Orthostatic hypotension is defined as ≥ 20 mm Hg reduction in systolic blood pressure and/or ≥ 10 mm Hg reduction in diastolic blood pressure between supine/semi-supine versus subsequent standing measurements.

   Note 2 (For Parkinson's Patients): If systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg, one repeat supine/semi-supine assessment is permitted within 5-10 minutes later, at the discretion of the PI (or delegate).
6. Heart rate in the range of 50 to 100 beats/minute after 5 minutes rest in supine/semi-supine position, and subsequently after 3 minutes of standing position.

Note: Participants with orthostatic hypotension are not permitted. Orthostatic hypotension is defined as ≥ 30 beats/minute increase in heart rate between supine/semi-supine versus subsequent standing measurements.

7. Body temperature (tympanic), between 35.5°C and 37.5°C. 8. Electrocardiogram (ECG) without clinically significant abnormal including QT interval corrected for Fredericia (QTcF) < 450 msec for male participants and < 470 msec for female participants.

9. No clinically significant findings in serum chemistry, haematology, coagulation or urinalysis (in the opinion of the Investigator).

10. Female participants must be of non-child-bearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone [FSH] level consistent with postmenopausal status, per local laboratory guidelines), or, if of child-bearing potential:

1. Must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test on Day -1, prior to dose administration.
2. Must agree not to donate ova or attempt to become pregnant from the time of signing consent until at least 30 days after the last dose of study drug.
3. If not exclusively in a same-sex relationship, must agree to remain abstinent throughout the study, or must agree to use adequate contraception (which is defined as use of a condom by the male partner combined with use of a highly effective method of contraception from one month prior to screening until at least 30 days after the last dose of study drug.

11. Male participants must:

1. Agree not to donate sperm from the time of signing consent until at least 30 days after the last dose of study drug.
2. If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as use of a condom plus a highly effective method of contraception from the time of signing consent until at least 30 days after the last dose of study drug.
3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, agree to use a condom from the time of signing consent until at least 30 days after the last dose of study drug.

12. Willing and able to comply with all scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria (Everyone)

Participants will be excluded from the study if there is evidence of any of the following:

1. Use of immunomodulators (including steroids and topical/oral/inhaled OTC glucocorticoids) within the past 60 days prior to the start of the first dose of study drug, unless approval is given by the study Sponsor (to be assessed at screening and Day -1)
2. Use of coenzyme Q10 within 5 days prior to the start of the first dose of study drug. (to be assessed at screening and Day -1)
3. Received a vaccine within 60 days of first dose of study drug (to be assessed at screening and Day -1)
4. History of hypersensitivity reaction, anaphylaxis or other clinically significant reactions or known allergy to any of the study drug ingredients.
5. History of transient ischemic attack or stroke or any unexplained loss of consciousness within 12 months of screening
6. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection upon admission to clinic on Day -1 (SARS-CoV-2 testing to be performed according to site standard process) or participant report of 'Long-COVID' any time prior to screening (where long-COVID is defined by probable or confirmed SARS-CoV-2 infection; usually within 3 months from the onset of COVID-19, with symptoms and effects that last for at least 2 months).
7. History of any clinically significant disorder (which, in the opinion of the Investigator [or delegate] would make implementation of the protocol or interpretation of study results difficult, or that would put the participant at risk by participating in the study), including cardiovascular (including but not limited to unstable angina, myocardial infarction, chronic heart failure), hematologic, pulmonary, hepatic, renal, gastrointestinal, connective tissue, uncontrolled endocrine/metabolic, oncologic (within the last 5 years excluding basal cell or squamous epithelial carcinomas of the skin that have been resected with clear margins and with no evidence of recurrence for at least 12 months), neurologic (including seizures, strokes, brain tumours), and psychiatric (including but not limited to major depression, schizophrenia, bipolar disorder, personality, or substance abuse disorder), or any disorder that may prevent the successful completion of the study or influence the absorption, distribution, metabolism, excretion, or action of the study drug.

   Note: Participants with well-controlled asthma (and is not receiving inhaled or oral steroids) is permitted, per PI (or delegate) discretion. Participants with well controlled, mild depression or anxiety, with no change in medication within the past 3 months is permitted, per PI (or delegate) discretion.
8. History of surgery or hospitalisation within 12 weeks prior to screening, or surgery planned during the study.
9. Lack of suitable veins for multiple venepunctures/cannulations as assessed by the Investigator or delegate at screening.
10. Presence of any tattoos or scarring which (in the opinion of the Investigator [or delegate]) would interfere with injection site reaction assessments.
11. Laboratory results at screening that indicate inadequate renal function (estimated creatinine clearance (CrCl) < 60mL/min (if either healthy and aged 40 and above or a Parkinson's patient) or < 79mL/min (if healthy and under 40 years)using the Cockcroft Gault formula).
12. Liver function test results elevated more than 1.5-fold above the ULN for gamma glutamyl transferase (GGT), alkaline phosphatase (ALP), aspartate aminotransferase (AST) or alanine aminotransferase (ALT). Volunteers with ALP and/or ALT/AST above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
13. Liver function tests outside the normal range for bilirubin (more than 1.5-fold above the ULN for total bilirubin).
14. Any clinically relevant laboratory finding or medical condition that could place the volunteer at risk for participation in the study.
15. Any active infection requiring systemic antibiotic, antifungal, or antiviral medication within 14 days prior to first dose of study drug (to be confirmed at screening and Day 1).
16. Concurrent enrolment in another clinical study, or participation in another clinical study within 90 days prior to screening.
17. Regular consumption of >10 standard alcoholic drinks/week where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc/Vol], 100 mL wine [12% Alc/Vol], 30 mL spirit [40% Alc/Vol]).
18. Positive alcohol breath or plasma test at screening or upon admission to the clinic on Day -1.
19. Positive urine drugs of abuse test at screening or upon admission to the clinic on Day -1.
20. Participant has a positive cotinine test upon admission to the clinic on Day -1.
21. Participant smokes more than 5 cigarettes or equivalent per week, and/or participant is unwilling to abstain from smoking for 72 hours prior to check-in on Day -1 and throughout the confinement period at the study site.
22. Use of cannabis or delta-9- tetrahydrocannabinol (THC), including for medicinal purposes, within 90 days prior to the start of the first dose of study drug, and/or participant is unwilling to abstain from use during the study
23. Participant is breastfeeding or pregnant, or planning to breastfeed or become pregnant during the study.
24. Known substance abuse or medical, psychological, or social conditions that, in the opinion of the PI (or delegate), may interfere with the participants inclusion in the clinical study or evaluation of the clinical study results.
25. Positive Hepatitis B surface antigen (HBsAg), Hepatitis C (HepC) virus antibody, or human immunodeficiency (HIV) antibody tests at screening.
26. Participant has donated blood/blood products, experienced significant (> 500 mL) blood loss within 3 months prior to the first dose administration or receipt of a blood transfusion within 1 year prior to the first dose administration.
27. Any other condition or prior therapy that in the opinion of the Investigator (or delegate) would make the participant unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Additional Inclusion Criteria (Parkinson's Disease Participants)

Parkinson's Disease Participants will be included in the study only if they satisfy all the following criteria:

1. Diagnosis of Parkinson's disease as defined by:

   • Evidence (written confirmation by a neurologist or geriatrician) of diagnosis of Parkinson's disease between 1-10 years prior to first dose administration.

   Note: Criteria for diagnosis of Parkinson's disease is per the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease:
   * Progressive asymmetric onset of bradykinesia
   * Muscle rigidity and/or rest tremor (4- to 6-Hz tremor in the fully resting limb)

     o Hoehn and Yahr score of 1-3 (inclusive)

     o Not diagnosed with any other neurodegenerative diseases.

     o If on levodopa containing medications: Stable levodopa containing medications for at least 2 months prior to screening with ability to be withdrawn from therapy for at least 12 hours (e.g., overnight) prior to study drug administration and on-study assessments. Participants will be able to resume therapy immediately after study drug is administrated and on-study assessments are completed.
     * If not on levodopa containing medications: To be able to remain treatment naïve throughout the study from screening through to the final EoS visit.

   Additional Exclusion Criteria (Parkinson's Disease Participants)

   Parkinson's Disease Participants will be excluded from the study if there is evidence of any of the following:

1. Use of antibiotics within 30 days prior to the start of the first dose of study drug (to be assessed at screening and Day -1).

2. Use of over-the-counter (OTC) prebiotics and probiotics supplements. Note: Participants receiving stable use of within 30 days prior to the start of the first dose of study drug may be permitted. (to be assessed at screening and Day -1).

3. History of use of any biologic therapy targeting beta-amyloid peptides or tau protein.

4. History of any brain surgery for Parkinson's disease, or a history of focused ultrasound treatment at any time, or history of any neuromodulation procedures.

5. Unexplained falls (≥ 3 falls) within 12 months prior to the start of the first dose of study drug.

6. History of in situ prostate carcinoma. 7. History of any concomitant disease, including cardiovascular (including but not limited to unstable angina, myocardial infarction, chronic heart failure), hematologic, pulmonary, hepatic, renal, gastrointestinal, connective tissue, uncontrolled endocrine/metabolic, neurologic (including seizures, strokes, brain tumours; but not including Parkinson's disease), and psychiatric (including but not limited to major depression, schizophrenia, bipolar disorder, personality, or substance abuse disorder), or any disorder that may prevent the successful completion of the study or influence the absorption, distribution, metabolism, excretion, or action of the study drug.

Note 1: Participants with diagnosed concomitant diseases that are considered stable by the PI for > 6 months (including those receiving stable concomitant therapy) may be permitted if agreed in consultation with the Sponsor.

Note 2: Participants with well-controlled asthma (and are not receiving inhaled or oral steroids) are permitted, per PI (or delegate) discretion.

1. Any history of cancer within the last 5 years (excluding basal cell or squamous epithelial carcinomas of the skin that have been resected with clear margins and with no evidence of recurrence for at least 12 months).
2. History of non-elective and/or non-routine surgery or hospitalisation within 12 weeks prior to screening, or surgery planned during the study, at the discretion of the PI.

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events [Safety and Tolerability] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  The peak plasma concentration of a drug after administration.
Elimination half life [T1/2] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  The time required for the concentration of the drug to reach half of its original value.
Time to reach Cmax [Tmax] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  Time required to reach Cmax.
Volume of Distribution [Vd] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  The apparent volume in which a drug is distributed (i.e., the parameter relating drug concentration in plasma to drug amount in the body).
Concentration [C] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  Amount of drug in a given volume of plasma
Area under the curve [AUC] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  The integral of the concentration-time curve (after a single dose or in steady state).
Clearance [CL] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  The volume of plasma cleared of the drug per unit time.
Bioavailability [f] | Day of treatment to end of follow-up period (1, 2 or 4 weeks)
  The systemically available fraction of a drug.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Alfred Hospital, Melbourne, Victoria
  - Nucleus Networks, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Michael J. Fox Trial Finder — https://www.michaeljfox.org/trial-finder
- See also: Shake It Up Trial Overview — https://shakeitup.org.au/longevity-trial/